CLINICAL TRIAL: NCT01607775
Title: Clinical Characterization of In-house Produced PMMA-cages in Patients With Cervical Pathology
Brief Title: In-house Produced PMMA- Versus PEEK-cages
Acronym: Palcage
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Universitätsmedizin Mannheim (Other)
Responsible Party: Principal Investigator, Martin Barth, MD, M. D., Vice-chairman, Universitätsmedizin Mannheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-256M-MA
Record Dates: First submitted 2012-05-22; First posted 2012-05-30 (Estimated); Last update posted 2012-06-05 (Estimated); Status verified 2012-06

CONDITIONS: Cervical Disc Degeneration; Cervical Stenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PEEK-cage (Active Comparator): Patients will receive a PEEK-cage
  Interventions: Device: Implantation of a PEEK-cage
- PMMA-cage (Experimental)
  Interventions: Device: PMMA-cage

INTERVENTIONS:
Device: Implantation of a PEEK-cage — A commercially avaliable cuboid cervical cage will be implantet
  Arms: PEEK-cage
Device: PMMA-cage — The in-house produced cervical cage will be implanted
  Arms: PMMA-cage

SUMMARY:
Subsidence of cervical cages is a common problem. For the study, a new polyacrylmethacrylate cage was designed and prospectively implanted in patients with a mono- or bilevel cervical pathology. As control, a commercially available PEEK-cage was used, patients were randomized using minimization randomization, controlling for age and bone mineral densitiy. The investigators hypothesize that the newly developed cage has similar clinical and radiological qualities compared to the PEEK-cage, but at a much more favourable cost-performance ratio.

ELIGIBILITY:
Inclusion Criteria:

* virgin spines
* no emergency operation
* age above 18
* sufficient knowledge of the German language
* indication for anterior cervical discectomy and fusion
* absence of concomitant spinal disease

Exclusion Criteria:

* prior cervical surgery
* indications other than ACDF
* concomitant neoplastic, metabolic, severe general or infectious disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2009-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
Clinical outcome (NDI) | 12 months postoperative
  NDI (Neck disability index) will be measured prior to surgery and 12 months after surgery. A difference of 20% between both groups is considered to be clinically significant, which is proposed for the experimental implant (PMMA-cage).

SECONDARY OUTCOMES:
Clinical outcome (VAS-neck), Subsidence | 12 months postoperative
  1. VAS-neck will be measured prior to surgery and 12 months after surgery. A difference of 20% between both groups is considered to be clinically significant, which is proposed for the experimental implant (PMMA-cage).
  2. Cage Subsidence will be measured using lateral radiographs prior to surgery and 12 months after surgery. Due to an improved cage design, significantly less subsidence is proposed for the experimental implant (PMMA-cage).